CLINICAL TRIAL: NCT02560311
Title: Long-term Outcome of HER2-amplified Metastatic Breast Cancer: A Retrospective Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr.2015-0050
Record Dates: First submitted 2015-09-02; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: ERBB2; Breast Cancer; Metastatic Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- HER2+ metastatic breast cancer
  Interventions: Other: observation

INTERVENTIONS:
Other: observation

SUMMARY:
The aim of this study is to analyze cases of human epidermal growth factor receptor (HER) 2-positive metastatic breast cancer (MBC) of the last 10 years at the University Hospital of Zurich to assess the efficacy of the treatment with trastuzumab in HER2-positive MBC and to find out associations between different variables and the outcome. The aim is to find out probable prognostic factors and patterns of disease progression. Prognostic factors could optimize treatment approaches and result in a delay of disease progression.

DETAILED DESCRIPTION:
Human epidermal growth factor (HER2) is a receptor tyrosine kinase and regulates diverse functions in normal cells such as growth, differentiation and survival of cells. In 25-30 per cent of breast cancer HER2 gene is amplified, what result in abnormally high levels of encoded HER2 protein in malignant cells. Overexpression or amplification of HER2 is associated with an aggressive form of breast cancer seen by significantly shortened disease-free survival and overall survival.

Trastuzumab, a humanized monoclonal antibody against the extracellular domain of HER2, inhibits the growth of breast tumor cells by receptor internalization, inhibition of cell-cycle progression and recruitment of immune-effector cells. Trastuzumab, as the first anti-HER2 therapy, is approved since 1998 in the United States and since 2000 in European countries for the treatment of HER2-overexpressing metastatic breast cancer (MBC). Single therapy as well as combination with chemotherapy has significantly improved the outcome of these women. Shown by longer time to disease progression, longer duration of response, lower rate of death at 1 year, longer survival and a 20 per cent reduction in the risk of death.

But still is little known about the long-term outcome nor patterns of disease progression of HER2-positive MBC. A few case reports showed a prolonged complete remission in HER2-positive MBC under an anti-HER2 treatment (trastuzumab, T-DM1, pertuzumab). These cases had some common characteristics such as negative hormone receptor status and metastasis to the live. Another hypothesis is a worse prognosis for patients with early development of CNS metastases.

ELIGIBILITY:
Inclusion Criteria:

* Received at least 1 dose of trastuzumab in metastatic setting at the University hospital of Zurich from 01/2004 to 12/2014.
* HER2+ status confirmed by immunohistochemistry (IHC) 3+ or fluorescence in situ hybridization (FISH) ≥ 2.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients with a human epidermal growth factor receptor (HER) 2+ breast cancer in metastatic stage (M1)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-09 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression | up to 120 months
  time from commencing trastuzumab (or other anti-HER2 therapy) to the time of disease progression or death

SECONDARY OUTCOMES:
Response duration | up to 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin J Dedes, Dr.med., Principal Investigator — UniversitätsSpital Zürich, Klinik für Gynäkologie; Bernhard Pestalozzi, Prof.Dr.med., Principal Investigator — UniversitätsSpital Zürich, Klinik für Onkologie
Locations (1):
- UniversitätsSpital Zürich, Klinik für Gynäkologie, Zurich, Canton of Zurich, Switzerland